CLINICAL TRIAL: NCT04889066
Title: A Phase II Clinical Trial of Durvalumab (MEDI4736) and Fractionated Stereotactic Radiotherapy (fSRT) Vs. Personalized Ultra-Fractionated Stereotactic Adaptive Radiotherapy (PULSAR) for the Treatment of Brain Metastases from Non-Small Cell Lung Cancer (NSCLC)
Brief Title: Durvalumab (MEDI4736) and Radiosurgery (fSRT Vs. PULSAR) for the Treatment of Non-Small Cell Lung Cancer Brain Metastases
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Project Never Initiated since sponsor stopped support for the trial- no human subjects were enrolled and no data regarding humans was collected or studied
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Principal Investigator, Kiran Kumar, Assistant Professor, University of Texas Southwestern Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STU-2021-0466
Record Dates: First submitted 2021-05-11; First posted 2021-05-17 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Brain Metastases from Non-small Cell Lung Cancer
Keywords: Non-small cell lung cancer; Immunotherapy; Durvalumab; Radiotherapy; PULSAR; Stereotactic ablative radiotherapy
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiosurgery; durvalumab

STUDY DESIGN:
Intervention Model Description: Based on investigator's hypothesis of improved rate of intracranial clinical benefit at 6-months from historical control of 60% to 86% and 10% attrition rate, a sample size of 23 patients is needed per study arm (total N=46) using a two-sided exact binomial test with a two-sided α=0.1 and power=80%.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Durvalumab and standard fSRT (Active Comparator): Fractionated stereotactic radiotherapy (fSRT) will be delivered to all previously untreated brain metastases noted at the time of treatment (up to 10 max). All brain metastases will be treated concurrently, 3 fractions total, delivered every other day (~2 times/week) with first cycle of Durvalumab.
  Interventions: Radiation: Stereotactic Radiation Therapy; Drug: Durvalumab
- Durvalumab and PULSAR (Experimental): Personalized ultra-fractionated stereotactic adaptive radiotherapy (PULSAR), will be delivered to all previously untreated brain metastases noted at the time of treatment (up to 10 max). All brain metastases will be treated concurrently, 3 "pulses" of radiation total, delivered one pulse monthly with each cycle of Durvalumab.
  Interventions: Radiation: Stereotactic Radiation Therapy; Drug: Durvalumab

INTERVENTIONS:
Radiation: Stereotactic Radiation Therapy — 24-27 Gy in 3 fractions- one plan, given once every other day with first cycle of Durvalumab for comparator arm. 24-27 Gy in 3 "pulses"- each pulse of radiation re-planned, given once every 4 weeks with each Durvalumab for experimental arm.
Drug: Durvalumab — Durvalumab (initially developed as MEDI4736) is a human monoclonal antibody of the immunoglobulin (Ig) G1 kappa subclass that inhibits binding of PD-L1 (B7-H1, CD274) to PD-1 (CD279) and CD80 (B7-1). MEDI4736 is composed of 2 identical heavy chains and 2 identical light chains, with an overall molecular weight of approximately 149 kDa. MEDI4736 contains a triple mutation in the constant domain of the Ig G1 heavy chain that reduces binding to complement protein C1q and the fragment crystallizable gamma receptors involved in triggering effector function.

SUMMARY:
This is a research study to find out if the new anti-cancer drug Durvalumab combined with radiation therapy to the brain will work in treating brain metastases from non-small cell lung cancer (NSCLC). Focused, highly precise radiation therapy to the brain, known as stereotactic radiosurgery (SRS), is a standard of care treatment that is commonly used for patients with metastatic lung cancer to the brain. It is standardly used as an alternative to surgery to eradicate the targeted tumours in the brain and prevent them from growing and causing symptoms. This study will look at the combination of the novel immunotherapy Durvalumab with two different ways of delivering SRS: 1) with each radiation treatment given every other day for 3 treatments with the first dose of Durvalumab (fSRT), or 2) with each radiation treatment, referred to as a "pulse," given every 4 weeks with each dose of Durvalumab for 3 treatments (PULSAR).

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven NSCLC primary with PD-L1 expression ≥ 1%
* At least one previously untreated, asymptomatic brain metastases (<=10 total) with at least one measurable (0.5 cm diameter or larger) as assessed by MRI
* No prior systemic treatment for metastatic NSCLC.
* age ≥ 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status 0 to 2
* Life expectancy greater than six (6) months
* Adequate normal organ and marrow function
* Body weight greater than 30 kg
* Ability to understand and willingness to sign written informed consent

Exclusion Criteria:

* Brain metastases that are symptomatic and/or with recent (<10 days) steroid use
* Active or prior documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]).
* Subjects may not be receiving any other investigational agents for the treatment of the cancer under study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, uncontrolled hypertension, unstable angina pectoris, cardiac arrhythmia, interstitial lung disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements, substantially increase risk of incurring AEs or compromise the ability of the patient to give written informed consent.
* Subjects must not be pregnant or nursing due to the potential for congenital abnormalities and the potential of this regimen to harm nursing infants.
* Administration of one or more lines of systemic therapy for the diagnosis of metastatic non-small cell lung cancer
* Prior receipt of systemic therapy for the management of high-risk early stage or locally advanced non-small cell lung cancer, prior to the development of metastatic disease, would not count towards the number of receipt of systemic therapy
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to durvalumab or other agents used in study
* Male or female patients of reproductive potential who are not willing to employ effective birth control from screening to 90 days after the last dose of durvalumab monotherapy
* Participation in another clinical study with an investigational product during the last 1 month
* Concurrent enrolment in another clinical study, unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study
* Receipt of the last dose of anticancer therapy (chemotherapy, immunotherapy, endocrine therapy, targeted therapy, biologic therapy, tumor embolization, monoclonal antibodies) ≤ 7 days prior to the first dose of study drug If sufficient wash-out time has not occurred due to the schedule or PK properties of an agent, a longer wash-out period will be required, as agreed by AstraZeneca and the investigator
* Any unresolved toxicity NCI CTCAE Grade ≥2 from previous anticancer therapy with the exception of alopecia, vitiligo, nausea, anorexia/weight loss, and the laboratory values defined in the inclusion criteria:

  * Patients with Grade ≥2 neuropathy will be evaluated on a case-by-case basis after consultation with the Study Physician.
  * Patients with irreversible toxicity not reasonably expected to be exacerbated by treatment with durvalumab may be included only after consultation with the Study Physician.
* Any other concurrent immunotherapy, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer-related conditions (e.g., hormone replacement therapy) is acceptable.
* Major surgical procedure (as defined by the Investigator) within 14 days prior to the first dose of immunotherapy.
* History of allogenic organ transplantation
* History of another primary malignancy except for:
* Malignancy treated with curative intent and with no known active disease ≥5 years before the first dose of immunotherapy and of low potential risk for recurrence
* Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
* Adequately treated carcinoma in situ without evidence of disease
* History of leptomeningeal carcinomatosis
* History of active primary immunodeficiency
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), hepatitis B (known positive HBV surface antigen (HBsAg) result), hepatitis C
* Current or prior use of immunosuppressive medication within 14 days before the first dose of durvalumab
* Receipt of live attenuated vaccine within 30 days prior to the first dose of immunotherapy
* Receipt of any prohibited medication

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-01 (Estimated); Study Completion 2025-01 (Estimated)

PRIMARY OUTCOMES:
Intercranial clinical benefit | 6 months after initiation of treatment
  Intracranial clinical benefit (Complete Response, Partial Response, or Stable Disease) assessed per the brain modified (bm) RECIST (response evaluation criteria in solid tumors) criteria

SECONDARY OUTCOMES:
Acute toxicity | 6- and 12-months after initiation of treatment
  All acute toxicities (CNS and non-CNS) will be evaluated using the NCI Common Terminology Criteria of Adverse Events (CTCAE) version 5.0, with results tabulated to examine frequency, severity, organs affected, and relationship to study treatment.
Quality of life questionnaire | 6- and 12-months after initiation of treatment
  Functional Assessment of Cancer Therapy brain (FACT-Br) questionnaires. scoring range 0-200. Higher the score, the better the QOL

CONTACTS AND LOCATIONS:
Overall Officials: Kiran Kumar, MD, Principal Investigator — University of Texas Southwestern Medical Center

IPD SHARING:
Plan to Share IPD: No